CLINICAL TRIAL: NCT03186235
Title: Regulatory T Cells and Their Cytokines Profile in Different Groups of Hepatitis c Infected Patients: A Case Control Study
Brief Title: T Regulatory Cells in Hepatitis c Infected Patients
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Hassan,MD, Principle Investigator, Assiut University
Other Study IDs: Esraa
Record Dates: First submitted 2017-06-10; First posted 2017-06-14 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group I : 18 healthy controls: Two milliliter of heparinized whole blood samples will be used for the Flow cytometry analysis to quantify percentages of circulating regulatory T cells in human peripheral blood in chronic hepatitis C patients in comparison with that of controls by four-colour flow cytometry analysis using a set of fluorochrome-labeled monoclonal antibodies against regulatory T cell surface markers and estimation of the level of IL35 by ElISA.
  Interventions: Other: Flow cytometry
- group II : 16 Hepatitis C infected patients (naïve): Two milliliter of heparinized whole blood samples will be used for the Flow cytometry analysis to quantify percentages of circulating regulatory T cells in human peripheral blood in chronic hepatitis C patients in comparison with that of controls by four-colour flow cytometry analysis using a set of fluorochrome-labeled monoclonal antibodies against regulatory T cell surface markers and estimation of the level of IL35 by ElISA.
  Interventions: Other: Flow cytometry
- group III:18 HCV-infected patients complicated with cirrhosis: Two milliliter of heparinized whole blood samples will be used for the Flow cytometry analysis to quantify percentages of circulating regulatory T cells in human peripheral blood in chronic hepatitis C patients in comparison with that of controls by four-colour flow cytometry analysis using a set of fluorochrome-labeled monoclonal antibodies against regulatory T cell surface markers and estimation of the level of IL35 by ElISA.
  Interventions: Other: Flow cytometry
- group IV: 18 HCV-infected patients with Hepatocellular cancer: Two milliliter of heparinized whole blood samples will be used for the Flow cytometry analysis to quantify percentages of circulating regulatory T cells in human peripheral blood in chronic hepatitis C patients in comparison with that of controls by four-colour flow cytometry analysis using a set of fluorochrome-labeled monoclonal antibodies against regulatory T cell surface markers and estimation of the level of IL35 by ElISA.
  Interventions: Other: Flow cytometry
- Group V:18 patients with sustained viral response (SVR).: Two milliliter of heparinized whole blood samples will be used for the Flow cytometry analysis to quantify percentages of circulating regulatory T cells in human peripheral blood in chronic hepatitis C patients in comparison with that of controls by four-colour flow cytometry analysis using a set of fluorochrome-labeled monoclonal antibodies against regulatory T cell surface markers and estimation of the level of IL35 by ElISA.
  Interventions: Other: Flow cytometry

INTERVENTIONS:
Other: Flow cytometry — Isolation of T regulatory cells from blood

SUMMARY:
Chronic hepatitis C infection is a global worldwide health problem with an increasing burden year-by-year, particularly in areas with a high endemicity like Egypt . The World Health Organization estimates that approximately 200 million people worldwide are infected with hepatitis c virus. In Egypt, it was estimated that 15 % of Egyptians have serologic evidence of hepatitis C viral infection .

DETAILED DESCRIPTION:
The ultimate outcome of hepatitis c viral infection is determined by the host immune response. Patients with acute hepatitis c viral infection who did not clear the virus developed chronicity. Persistant hepatitis c virus -specific cytotoxic T-cell responses in the liver have been associated with the development of hepatic inflammation which may ultimately lead to liver cirrhosis. One of the potential mechanisms that might modulate hepatitis c virus -specific immune responses is the inhibitory role of the regulatory T cells.

Regulatory T cells are a subtype of T-cells that play a fundamental role in maintaining immune homeostasis to balance between the tissue-damaging and protective effects of the immune response. Regulatory T cells are characterized by the expression of the Forkhead box protein P3 transcription factor in the nucleus and is generally accepted as the single best marker for regulatory Tcells. In cases of hepatitis c virus infection, the role of regulatory Tcells is still controversial and most of studies yielded conflicting reports. This conflict may be explained by the heterogeneity in the methods and sites of studying the frequency of regulatory T cells.

There are strong evidences that regulatory T cells and their cytokines may play an important role in the induction of tolerance in the liver.

Interleukin 35 is an immune-suppressive cytokine expressed in stimulated human regulatory Tcells during inflammatory responses and consists of Interlukin-12a ( Interleukin 12p35 subunit) and IL-27b chains, encoded by the Interleukin 12A and Epstien Bar I3 genes, respectively. It is a novel heterodimeric cytokine belonging to the Interleukin 12 family, and little is known about its receptor. Activated peripheral blood mononuclear cell (PBMC)- derived human regulatory T cells have been shown to express and secrete large amounts of Interleukin 35, which contributes significantly to the suppressive capacity of regulatory T cells in an Interlukin 35-dependent manner.

Additionally, human regulatory T cell -derived IL35 is required for the conversion of human conventional cluster of differentiation 4+Foxp3_ T cells into induced T regulatory 35 cells, which then promote the generation of more induced T regulatory 35 cells via Interleukin 35 secretion, resulting in infectious tolerance (18). In addition, Interleukin 35 has been shown to suppress the T helper (Th) cells Th1 and Th17.

In this study, investigators will evaluate the possible role of regulatory T cells and their cytokines in different groups of hepatitis c infected patients by investigating the frequency of regulatory T cells and serum level of IL35 and examining their relationship to the various patterns of hepatitis c viral persistence, hepatitis c virus pathogenesis, complications with cirrhosis and hepatocellular carcinoma in an attempt to estimate the future value of using anti IL35 and regulatory T cell depletion in those patients.

ELIGIBILITY:
Inclusion Criteria:

* positive for hepatitis c viral antibodies by Enzyme Linked Immuno Sorbent Assay and by hepatitis c viral Ribo Nucleic Acid Real time Polymerase Chain Reaction

Exclusion Criteria:

* are pregnancy, history of Schistosoma infection, inflammatory bowel diseases or suspected inflammatory bowel diseases , autoimmune diseases including rheumatoid arthritis, and any patients on systemic immunomodulators

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: . All participants were recruited from Assiut Liver Institute for Treatment of Hepatitis C Virus and Assiut University Hospitals outpatient clinics, Assiut, Egypt. Healthy donors will be attending blood bank of Assiut University Hospital during the study period. They will be negative for known serologic markers of hepatitis (B & C) including hepatitis B surface antigen and antibodies to Hepatitis C virus
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
frequency of T regulatory cells in all 6 groups using flow cytometry | An average 1 year
  frequency of T regulatory cells will be estimated by flow cytometry in all 6 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lauer GM, Walker BD. Hepatitis C virus infection. N Engl J Med. 2001 Jul 5;345(1):41-52. doi: 10.1056/NEJM200107053450107. No abstract available. PMID 11439948
- [Background] Klenerman P, Thimme R. T cell responses in hepatitis C: the good, the bad and the unconventional. Gut. 2012 Aug;61(8):1226-34. doi: 10.1136/gutjnl-2011-300620. Epub 2011 Aug 28. PMID 21873736
- [Background] Bowen DG, Walker CM. Adaptive immune responses in acute and chronic hepatitis C virus infection. Nature. 2005 Aug 18;436(7053):946-52. doi: 10.1038/nature04079. PMID 16107834
- [Background] Hartling HJ, Gaardbo JC, Ronit A, Knudsen LS, Ullum H, Vainer B, Clausen MR, Skogstrand K, Gerstoft J, Nielsen SD. CD4(+) and CD8(+) regulatory T cells (Tregs) are elevated and display an active phenotype in patients with chronic HCV mono-infection and HIV/HCV co-infection. Scand J Immunol. 2012 Sep;76(3):294-305. doi: 10.1111/j.1365-3083.2012.02725.x. PMID 22671952
- [Background] Sturm N, Thelu MA, Camous X, Dimitrov G, Ramzan M, Dufeu-Duchesne T, Bonorino P, Guillermet C, Brambilla E, Arvers P, Pernollet M, Leroy V, Zarski JP, Marche PN, Jouvin-Marche E. Characterization and role of intra-hepatic regulatory T cells in chronic hepatitis C pathogenesis. J Hepatol. 2010 Jul;53(1):25-35. doi: 10.1016/j.jhep.2010.02.024. Epub 2010 Apr 20. PMID 20452085
- [Background] Sakaguchi S, Yamaguchi T, Nomura T, Ono M. Regulatory T cells and immune tolerance. Cell. 2008 May 30;133(5):775-87. doi: 10.1016/j.cell.2008.05.009. PMID 18510923
- [Background] Magg T, Mannert J, Ellwart JW, Schmid I, Albert MH. Subcellular localization of FOXP3 in human regulatory and nonregulatory T cells. Eur J Immunol. 2012 Jun;42(6):1627-38. doi: 10.1002/eji.201141838. PMID 22678915
- [Background] Adams DH, Eksteen B, Curbishley SM. Immunology of the gut and liver: a love/hate relationship. Gut. 2008 Jun;57(6):838-48. doi: 10.1136/gut.2007.122168. Epub 2008 Jan 18. No abstract available. PMID 18203807